CLINICAL TRIAL: NCT03860441
Title: Holistic Approach for Active and Healthy Aging: Physical and Cognitive Activity, and Nutrition
Brief Title: Effects of Cognitive Intervention on Cognition, Mobility and Brain Electrocortical Activity
Acronym: GIBKOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Science and Research Centre Koper (Other)
Collaborators: University of Primorska (Other); Albert Einstein College of Medicine (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GIBKOP2017
Record Dates: First submitted 2018-10-02; First posted 2019-03-04 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Cognitive Decline; Cognitive Impairment; Aging; Motor Coordination or Function
Keywords: cognition; mobility; cognitive reserve; EEG/ERP
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Remediation; Cognitive Training

STUDY DESIGN:
Intervention Model Description: Participants in the intervention group followed a computerized cognitive training program for 2-months, 3x/week, 40min/session
Who Masked: Participant
Masking Description: A single-blind randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group received 24 sessions of computerized cognitive training, with a total time of 960 min.
  Interventions: Other: Computerized cognitive training
- Active control group (Active Comparator): Participants in the control group attended activities separate activities, such as learning about healthy lifestyle, had cooking and other social lessons for the same amount as the intervention group performed cognitive training.
  Interventions: Other: Computerized cognitive training

INTERVENTIONS:
Other: Computerized cognitive training — Intervention used CogniFit platform with Personalized brain training sub-option
  Other Names: cognitive remediation; cognitive training

SUMMARY:
Within this project the investigators tested the effectiveness of 2-month of computerized cognitive training (CCT) on CogniFit online platform on 77 older adults, which were randomly divided into intervention and control group. The investigators tested close (battery of cognitive functions) and far transfer (postural and mobility control, EEG, blood samples) of the CCT. Additionally, the investigators were interested into seeing a long-lasting effect, therefore participants were brought back to the laboratory 1 year post CCT.

ELIGIBILITY:
Inclusion Criteria:

* active and healthy older adults with no major health issues
* members of the Center for Daily Activity Koper (Slovenia)
* had normal or corrected-to-normal vision;
* reported no history of cardiovascular, neurological, or psychiatric conditions

Exclusion Criteria:

* younger than 60
* smoking; regular alcohol consumption;
* acute or chronic skeletal, neuromuscular, metabolic and cardiovascular disease condition;

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change in gait speed | up to 8 weeks
  The primary outcome is change in gait speed during single- and dual-task conditions from baseline to post-intervention.

SECONDARY OUTCOMES:
Executive control (Trail-Making Task Forms A and B) | up to 8 weeks
  Secondary outcome is change in executive control, measured with TMT A and B tests
Sensorimotor integration measured with EEG/ERP methodology | up to 8 weeks
  Secondary outcome is change ERP components P1, N1, P2 and P3 (amplitudes and latencies)
Brain-derived neurotrophic factor (BDNF) extracted from peripheral blood sampling | up to 8 weeks
  Secondary outcome is change in plasma BDNF plasma extraction evaluated in pg/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Daily Activity Koper (Slovenia), Koper, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marusic U, Kavcic V, Giordani B, Gerzevic M, Meeusen R, Pisot R. Computerized spatial navigation training during 14 days of bed rest in healthy older adult men: Effect on gait performance. Psychol Aging. 2015 Jun;30(2):334-340. doi: 10.1037/pag0000021. Epub 2015 May 4. PMID 25938245
- [Result] Verghese J, Mahoney J, Ambrose AF, Wang C, Holtzer R. Effect of cognitive remediation on gait in sedentary seniors. J Gerontol A Biol Sci Med Sci. 2010 Dec;65(12):1338-43. doi: 10.1093/gerona/glq127. Epub 2010 Jul 19. PMID 20643703
- [Result] Marusic U, Verghese J, Mahoney JR. Cognitive-Based Interventions to Improve Mobility: A Systematic Review and Meta-analysis. J Am Med Dir Assoc. 2018 Jun;19(6):484-491.e3. doi: 10.1016/j.jamda.2018.02.002. Epub 2018 Apr 19. PMID 29680203